CLINICAL TRIAL: NCT03154190
Title: St. Judes-Stanford Comprehensive Support Initiative
Brief Title: Health Care Coach Support in Reducing Acute Care Use and Cost in Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Manali Indravadan Patel, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: VAR0134
Record Dates: First submitted 2016-11-14; First posted 2017-05-16 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Acute Myeloid Leukemia; Brain Glioblastoma; Estrogen Receptor Negative; Extensive Stage Small Cell Lung Carcinoma; Head and Neck Carcinoma; HER2/Neu Negative; Hormone-Resistant Prostate Cancer; Limited Stage Small Cell Lung Carcinoma; Myelodysplastic Syndrome; Progesterone Receptor Negative; Progressive Disease; Recurrent Carcinoma; Stage II Pancreatic Cancer; Stage II Rectal Cancer; Stage IIA Pancreatic Cancer; Stage IIA Rectal Cancer; Stage IIB Pancreatic Cancer; Stage IIB Rectal Cancer; Stage IIC Rectal Cancer; Stage III Colon Cancer; Stage III Esophageal Cancer; Stage III Gastric Cancer; Stage III Non-Small Cell Lung Cancer; Stage III Ovarian Cancer; Stage III Pancreatic Cancer; Stage III Rectal Cancer; Stage III Skin Melanoma; Stage IIIA Colon Cancer; Stage IIIA Esophageal Cancer; Stage IIIA Gastric Cancer; Stage IIIA Non-Small Cell Lung Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Rectal Cancer; Stage IIIA Skin Melanoma; Stage IIIB Colon Cancer; Stage IIIB Esophageal Cancer; Stage IIIB Gastric Cancer; Stage IIIB Non-Small Cell Lung Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Rectal Cancer; Stage IIIB Skin Melanoma; Stage IIIC Colon Cancer; Stage IIIC Esophageal Cancer; Stage IIIC Gastric Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Rectal Cancer; Stage IIIC Skin Melanoma; Stage IV Bladder Cancer; Stage IV Bone Sarcoma; Stage IV Breast Cancer; Stage IV Colon Cancer; Stage IV Esophageal Cancer; Stage IV Gastric Cancer; Stage IV Non-Small Cell Lung Cancer; Stage IV Ovarian Cancer; Stage IV Pancreatic Cancer; Stage IV Rectal Cancer; Stage IV Renal Cell Cancer; Stage IV Skin Melanoma; Stage IV Soft Tissue Sarcoma; Stage IVA Bone Sarcoma; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Bone Sarcoma; Stage IVB Colon Cancer; Stage IVB Rectal Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Disease Progression; Recurrence; Pancreatic Neoplasms; Rectal Neoplasms; Colonic Neoplasms; Esophageal Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Ovarian Neoplasms; Melanoma; Urinary Bladder Neoplasms; Bone Neoplasms; Breast Neoplasms; Carcinoma, Renal Cell; Sarcoma; Triple Negative Breast Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (usual care) (Active Comparator): Patients receive usual care.
  Interventions: Other: Best Practice; Other: Laboratory Biomarker Analysis; Other: Survey Administration
- Arm B (health care coach support) (Experimental): Patients undergo health care coach support with a baseline introduction (either telephonic or in-person) of the program followed by a visit (telephonic or in-person) with the health care coach after the first oncology appointment to discuss goals of care. The health care coach will contact patient based on patients' ongoing needs (weekly to monthly) and will conduct symptom assessments based on patients' treatment plans and symptoms.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Supportive Care; Other: Survey Administration

INTERVENTIONS:
Other: Best Practice — Receive usual care
  Other Names: standard of care; standard therapy
  Arms: Arm A (usual care)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Supportive Care — Undergo health care coach support
  Other Names: Supportive Therapy; Symptom Management; Therapy, Supportive
  Arms: Arm B (health care coach support)
Other: Survey Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies health care coach support in reducing acute care use and cost in patients with cancer. Health care coach support may help cancer patients to make decisions about their care that matches what is important to them with symptom management.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To reduce acute care utilization by 2-5% for advanced cancer patients by training and deploying health care coaches who help patients and families discuss care goals, virtual modalities, engage in shared-decision-making, and participate in educational activities.

SECONDARY OBJECTIVES:

I. To improve patients' experience of their care. II. Improve patient understanding of advanced care planning. III. To improve the receipt of goal concordant care. IV. To reduce total healthcare costs.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive usual care.

ARM B: Patients undergo health care coach support with a baseline introduction (either telephonic or in-person) of the program followed by a visit (telephonic or in-person) with the health care coach after the first oncology appointment to discuss goals of care. The health care coach will contact patient based on patients' ongoing needs (weekly to monthly) and will conduct symptom assessments based on patients' treatment plans and symptoms.

After completion of study, patients are followed up for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed patients for the following conditions

  * Colon cancer stage III and IV
  * Rectal cancer stage II, III, IV
  * Glioblastoma multiforme (brain) -- no stage
  * Non-small cell lung cancer stage IIIA, IIIB, IV
  * Small cell lung cancer, limited stage and extensive stage
  * Castration-resistant prostate cancer
  * Head and neck cancer stage III and IV
  * Gastric cancer stage III and IV
  * Esophageal cancer stage III and IV
  * Pancreatic cancer stage II, III, IV
  * Renal cell carcinoma, stage IV
  * Breast cancer, stage IV, if triple negative ER/PR/H2N negative or on systemic chemotherapy
  * Sarcoma, stage IV
  * Bladder carcinoma, stage IV
  * Acute myeloid leukemia
  * Melanoma, stage III and IV
  * Ovarian cancer, stage III and IV
  * High grade myelodysplastic syndrome (MDS)
* Any patient with recurrent or progressive cancer
* Patients must have the ability to understand and willingness to sign a written informed consent document
* Patient must have ongoing oncologic needs and plan to receive all care at the study institution and not already be in hospice or home-care

Exclusion Criteria:

* Patients must have capacity to consent
* Pregnant patients are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manali Patel, Principal Investigator — Stanford University
Locations (1):
- Virginia K Crosson Cancer Center, Fullerton, California, United States

REFERENCES:
- [Derived] Patel MI, Kapphahn K, Dewland M, Aguilar V, Sanchez B, Sisay E, Murillo A, Smith K, Park DJ. Effect of a Community Health Worker Intervention on Acute Care Use, Advance Care Planning, and Patient-Reported Outcomes Among Adults With Advanced Stages of Cancer: A Randomized Clinical Trial. JAMA Oncol. 2022 Aug 1;8(8):1139-1148. doi: 10.1001/jamaoncol.2022.1997. PMID 35771552
- [Derived] Patel MI, Aguilar V, Sanchez B, Sisay E, Park DJ. Health care coach support to assist with advance care planning and symptom management -A randomized controlled trial. Contemp Clin Trials. 2021 Dec;111:106617. doi: 10.1016/j.cct.2021.106617. Epub 2021 Nov 5. PMID 34749008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Started | 64 | 64
6 Months | 41 | 44
Completed | 30 | 28
Not Completed | 34 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support) | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Median (Full Range); unit: years] | 67 [43 to 89] | 70 [19 to 89] | 67 [19 to 89]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Female | 31 | 30 | 61
  Gender Identity: Male | 32 | 32 | 64
  Gender Identity: Non-binary | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 12 | 23
  Not Hispanic or Latino | 53 | 52 | 105
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 7 | 4 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 2 | 5
  White | 40 | 46 | 86
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 10 | 10 | 20
Education Level [Count of Participants; unit: Participants]
  Less than 8th Grade | 1 | 0 | 1
  Some High School | 1 | 1 | 2
  High School Graduate or GED | 5 | 8 | 13
  4-Year College Graduate | 11 | 8 | 19
  Some College or 2-Year Degree | 22 | 20 | 42
  More than 4-Year College Graduate | 6 | 14 | 20
  Prefer Not To Answer | 18 | 13 | 31
Insurance Status [Count of Participants; unit: Participants]
  Medicare | 20 | 21 | 41
  Medicaid | 3 | 3 | 6
  Private | 40 | 38 | 78
  Uninsured | 1 | 2 | 3
Anatomic Site of Cancer Diagnosis [Count of Participants; unit: Participants]
  Gynecology | 4 | 7 | 11
  Genitourinary | 3 | 5 | 8
  Gastrointestinal | 29 | 20 | 49
  Breast | 5 | 4 | 9
  Thoracic | 10 | 14 | 24
  Malignant Hematologic | 5 | 5 | 10
  Head and Neck | 1 | 5 | 6
  Melanoma | 2 | 2 | 4
  Glioblastoma | 4 | 2 | 6
  Unknown Primary | 1 | 0 | 1
Cancer Stage at Diagnosis [Count of Participants; unit: Participants]
  3 | 9 | 12 | 21
  4 | 49 | 48 | 97
  Not applicable (i.e., Leukemia, Glioblastoma) | 6 | 4 | 10
Cancer-Directed Treatment [Number; unit: participants]
  Chemotherapy | 60 | 60 | 120
  Radiation | 28 | 25 | 53
  Surgery | 10 | 19 | 29
Recurrent Cancer - no [Count of Participants; unit: Participants] | 29 | 23 | 52
Symptom Burden [Mean (Standard Deviation); unit: score on a scale] — Symptom-burden was assessed by summing 10 items of the Edmonton Assessment Scale (0-10) resulting in a range from 0-100. Lower scores indicate better symptom control, while higher scores indicated worse symptoms by patients with cancer.
  score on a scale | 12.8 (11.5) | 13.3 (10.5) | 13 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Emergency Department Visits (Chart Review)
Description: Mean emergency department visits for each patient will be abstracted by electronic medical record chart review for each patient at 6 months after enrollment. We will evaluate comparisons of mean numbers of emergency department visits between study arms.
Time Frame: 6 months after patient enrollment
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
visits | 1.33 (2.53) | 0.41 (1.02)
Statistical Analysis 1: Comparison: Arm A (Usual Care) vs Arm B (Health Care Coach Support); Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.30, 95% CI 2-sided [0.20 to 0.47]

2. Primary Outcome: Number of Hospitalization Visits (Chart Review)
Description: Mean Hospitalization use for each patient will be abstracted by electronic medical record chart review for each patient at 6 months after enrollment. We will evaluate comparisons of mean numbers of hospitalizations between the two study arms.
Time Frame: 6 months after patient enrollment
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
visits | 0.91 (1.98) | 0.44 (1.28)
Statistical Analysis 1: Comparison: Arm A (Usual Care) vs Arm B (Health Care Coach Support); Test type: Superiority; Regression, Cox; Hazard Ratio (HR) = 0.48, 95% CI 2-sided [0.30 to 0.75]

3. Secondary Outcome: Change in Patient Satisfaction With Care and Decision Making Among Patients Undergoing Health Care Coach Support as Assessed by Consumer Assessment of Healthcare Providers and Systems-G and Patient Satisfaction With Decision Scale
Description: Each patient will receive a satisfaction with decision-making survey (The Satisfaction with Decision Survey) at baseline, 6 months, and 12 months.
  Satisfaction with Decision was assessed using the Satisfaction with Decision scale, which measured rating of decision-making. Questions were assessed with responses on a scale of "strongly disagree," "disagree," "neither agree nor disagree," "agree," or "strongly agree." Results are expressed as proportion of participants who responded "strongly agree."
Time Frame: Change in patient satisfaction with care and decision making from baseline to 6 and 12 months
Population: Participants who completed the survey at each respective time point are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 47 | 51
Participants
  Baseline: I am satisfied that I am adequately informed about the treatment decisions available to me | 47 | 50
  6 Month: I am satisfied that I am adequately informed about the treatment decisions available to me: number analyzed (Participants) | 41 | 44
  6 Month: I am satisfied that I am adequately informed about the treatment decisions available to me | 40 | 44
  12 Month: I am satisfied that I am adequately informed about the treatment decisions available to me: number analyzed (Participants) | 30 | 28
  12 Month: I am satisfied that I am adequately informed about the treatment decisions available to me | 29 | 28
  Baseline: I made the best decisions possible about my treatment options | 47 | 50
  6 Month: I made the best decisions possible about my treatment options: number analyzed (Participants) | 41 | 44
  6 Month: I made the best decisions possible about my treatment options | 40 | 44
  12 Month: I made the best decisions possible about my treatment options: number analyzed (Participants) | 30 | 28
  12 Month: I made the best decisions possible about my treatment options | 29 | 28
  Baseline: I believe that my decisions were consistent with what's important to me | 47 | 50
  6 Month: I believe that my decisions were consistent with what's important to me: number analyzed (Participants) | 41 | 44
  6 Month: I believe that my decisions were consistent with what's important to me | 40 | 44
  12 Month: I believe that my decisions were consistent with what's important to me: number analyzed (Participants) | 30 | 28
  12 Month: I believe that my decisions were consistent with what's important to me | 29 | 28
  Baseline: I expect to successfully carry out (or continue to carry out) the decision I made | 47 | 50
  6 Month: I expect to successfully carry out (or continue to carry out) the decision I made: number analyzed (Participants) | 41 | 44
  6 Month: I expect to successfully carry out (or continue to carry out) the decision I made | 40 | 44
  12 Month: I expect to successfully carry out (or continue to carry out) the decision I made: number analyzed (Participants) | 30 | 28
  12 Month: I expect to successfully carry out (or continue to carry out) the decision I made | 29 | 28
  Baseline: I was encouraged by the Cancer Center staff to speak up about my treatment preferences | 47 | 50
  6 Month: I was encouraged by the Cancer Center staff to speak up about my treatment preferences: number analyzed (Participants) | 41 | 44
  6 Month: I was encouraged by the Cancer Center staff to speak up about my treatment preferences | 40 | 44
  12 Month: I was encouraged by the Cancer Center staff to speak up about my treatment preferences: number analyzed (Participants) | 30 | 28
  12 Month: I was encouraged by the Cancer Center staff to speak up about my treatment preferences | 29 | 28
  Baseline: I am satisfied with the care I received at St. Joseph Heritage Healthcare | 46 | 50
  6 Month: I am satisfied with the care I received at St. Joseph Heritage Healthcare: number analyzed (Participants) | 41 | 44
  6 Month: I am satisfied with the care I received at St. Joseph Heritage Healthcare | 39 | 44
  12 Month: I am satisfied with the care I received at St. Joseph Heritage Healthcare: number analyzed (Participants) | 30 | 28
  12 Month: I am satisfied with the care I received at St. Joseph Heritage Healthcare | 28 | 28

4. Secondary Outcome: Change in Patient Satisfaction With Care Among Patients Undergoing Health Care Coach Support as Assessed by Consumer Assessment of Healthcare Providers and Systems-G.
Description: Each patient will receive a satisfaction with care survey (The Consumer Assessment of Healthcare Providers and Systems-G) at baseline, 6 months, and 12 months.
  Overall Health and Overall Mental or Emotional health was assessed using the Consumer Assessment of Health Care Providers and Systems-Clinician and Group Survey version 2.0 (cite) questions #26, which measured rating of overall health with responses, "excellent," "very good," "fair," or "poor." Questions were assessed with responses "never", "sometimes," "usually," or "always," or care rated as "worst," "fair," good", or "best." Results are expressed as proportion of participants who responded "always", or "best care."
Time Frame: Change in patient satisfaction with care from baseline to 6 and 12 months
Population: Participants who completed the survey at each respective time point are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 47 | 64
Participants
  Baseline: How often did you get an answer to your medical question the same day during office hours?: number analyzed (Participants) | 28 | 32
  Baseline: How often did you get an answer to your medical question the same day during office hours? | 22 | 22
  6 Month: How often did you get an answer to your medical question the same day during office hours?: number analyzed (Participants) | 27 | 34
  6 Month: How often did you get an answer to your medical question the same day during office hours? | 21 | 34
  12 Month: How often did you get an answer to your medical question the same day during office hours?: number analyzed (Participants) | 20 | 21
  12 Month: How often did you get an answer to your medical question the same day during office hours? | 15 | 17
  Baseline: How often did you get an answer to your medical question the same day after office hours?: number analyzed (Participants) | 18 | 12
  Baseline: How often did you get an answer to your medical question the same day after office hours? | 11 | 9
  6 Month: How often did you get an answer to your medical question the same day after office hours?: number analyzed (Participants) | 13 | 13
  6 Month: How often did you get an answer to your medical question the same day after office hours? | 9 | 13
  12 Month : How often did you get an answer to your medical question the same day after office hours?: number analyzed (Participants) | 8 | 11
  12 Month : How often did you get an answer to your medical question the same day after office hours? | 6 | 10
  Baseline: How often did your provider team explain things in a way that was easy to understand?: number analyzed (Participants) | 47 | 51
  Baseline: How often did your provider team explain things in a way that was easy to understand? | 34 | 38
  6 Month : How often did your provider team explain things in a way that was easy to understand?: number analyzed (Participants) | 41 | 44
  6 Month : How often did your provider team explain things in a way that was easy to understand? | 35 | 42
  12 Month: How often did your provider team explain things in a way that was easy to understand?: number analyzed (Participants) | 29 | 28
  12 Month: How often did your provider team explain things in a way that was easy to understand? | 27 | 24
  Baseline: How often did this provider's team listen carefully to you?: number analyzed (Participants) | 47 | 51
  Baseline: How often did this provider's team listen carefully to you? | 40 | 46
  6 Month: How often did this provider's team listen carefully to you?: number analyzed (Participants) | 41 | 44
  6 Month: How often did this provider's team listen carefully to you? | 37 | 42
  12 Month: How often did this provider's team listen carefully to you?: number analyzed (Participants) | 30 | 28
  12 Month: How often did this provider's team listen carefully to you? | 28 | 26
  Baseline: How often did this provider's team show respect for what you had to say?: number analyzed (Participants) | 47 | 51
  Baseline: How often did this provider's team show respect for what you had to say? | 42 | 47
  6 Month: How often did this provider's team show respect for what you had to say?: number analyzed (Participants) | 41 | 44
  6 Month: How often did this provider's team show respect for what you had to say? | 38 | 43
  12 Month: How often did this provider's team show respect for what you had to say?: number analyzed (Participants) | 30 | 64
  12 Month: How often did this provider's team show respect for what you had to say? | 30 | 28
  Baseline: How often did this provider's team spend enough time with you?: number analyzed (Participants) | 46 | 51
  Baseline: How often did this provider's team spend enough time with you? | 40 | 41
  6 Month: How often did this provider's team spend enough time with you?: number analyzed (Participants) | 41 | 44
  6 Month: How often did this provider's team spend enough time with you? | 40 | 44
  12 Month: How often did this provider's team spend enough time with you?: number analyzed (Participants) | 30 | 28
  12 Month: How often did this provider's team spend enough time with you? | 30 | 28
  Baseline: How often did your provider's office follow up to give you the results of a test?: number analyzed (Participants) | 43 | 50
  Baseline: How often did your provider's office follow up to give you the results of a test? | 37 | 39
  6 Month: How often did your provider's office follow up to give you the results of a test?: number analyzed (Participants) | 39 | 44
  6 Month: How often did your provider's office follow up to give you the results of a test? | 35 | 38
  12 Month: How often did your provider's office follow up to give you the results of a test?: number analyzed (Participants) | 30 | 28
  12 Month: How often did your provider's office follow up to give you the results of a test? | 28 | 24
  Baseline: I am satisfied with the care I received at St. Joseph Heritage Health Care?: number analyzed (Participants) | 47 | 51
  Baseline: I am satisfied with the care I received at St. Joseph Heritage Health Care? | 47 | 50
  6 Month: I am satisfied with the care I received at St. Joseph Heritage Health Care?: number analyzed (Participants) | 41 | 44
  6 Month: I am satisfied with the care I received at St. Joseph Heritage Health Care? | 40 | 44
  12 Month: I am satisfied with the care I received at St. Joseph Heritage Health Care?: number analyzed (Participants) | 30 | 28
  12 Month: I am satisfied with the care I received at St. Joseph Heritage Health Care? | 27 | 28
  Baseline: Received the best care?: number analyzed (Participants) | 46 | 52
  Baseline: Received the best care? | 30 | 37
  6 Month: Received the best care?: number analyzed (Participants) | 41 | 44
  6 Month: Received the best care? | 27 | 33
  12 Month: Received the best care?: number analyzed (Participants) | 30 | 28
  12 Month: Received the best care? | 21 | 22
  Baseline: In general, how would you rate your overall health?: number analyzed (Participants) | 46 | 52
  Baseline: In general, how would you rate your overall health? | 12 | 12
  6 Month: In general, how would you rate your overall health?: number analyzed (Participants) | 41 | 44
  6 Month: In general, how would you rate your overall health? | 10 | 12
  12 Month: In general, how would you rate your overall health?: number analyzed (Participants) | 30 | 28
  12 Month: In general, how would you rate your overall health? | 9 | 9
  Baseline: In general, how would you rate your overall mental or emotional health?: number analyzed (Participants) | 46 | 52
  Baseline: In general, how would you rate your overall mental or emotional health? | 31 | 34
  6 Month: In general, how would you rate your overall mental or emotional health?: number analyzed (Participants) | 41 | 44
  6 Month: In general, how would you rate your overall mental or emotional health? | 13 | 28
  12 Month: In general, how would you rate your overall mental or emotional health?: number analyzed (Participants) | 31 | 29
  12 Month: In general, how would you rate your overall mental or emotional health? | 9 | 18

5. Secondary Outcome: Mean Emergency Department Visits (Chart Review)
Description: Emergency Department use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of emergency department visits between study arms.
Time Frame: 12 months after patient enrollment
Measure: Mean (Standard Deviation); unit: mean visits per year
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
mean visits per year | 2.02 (3.86) | 0.92 (1.67)
Statistical Analysis 1: Comparison: Arm A (Usual Care) vs Arm B (Health Care Coach Support); Test type: Superiority; Risk Ratio (RR) = 0.45, 95% CI 2-sided [0.33 to 0.62]

6. Secondary Outcome: Number of People With Emergency Department Visit (Chart Review)
Description: Number of people with Emergency Department use in the 30 days before death will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of the number of people with emergency department visits between study arms.
Time Frame: 30 days prior to death
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 26 | 32
Participants | 4 | 0

7. Secondary Outcome: Hospitalization Visits (Chart Review)
Description: Hospital use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of hospitalization use between study arms.
Time Frame: 12 months after patient enrollment
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
visits | 1.63 (3.03) | 0.82 (1.68)
Statistical Analysis 1: Comparison: Arm A (Usual Care) vs Arm B (Health Care Coach Support); Test type: Superiority; Risk Ratio (RR) = 0.50, 95% CI 2-sided [0.36 to 0.70]

8. Secondary Outcome: Number of Patients With Hospital Use (Chart Review)
Description: Number of patients with hospital use in the 30 days before death will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of proportion of people with hospitalization use between study arms in the 30 days before death.
Time Frame: 30 days prior to death
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 26 | 32
Participants | 3 | 0

9. Secondary Outcome: Hospice Consult (Chart Review)
Description: Hospice use for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of hospice use between study arms.
Time Frame: 6 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
Participants | 10 | 20

10. Secondary Outcome: Hospice Consult (Chart Review)
Description: as for outcome 9
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
Participants | 10 | 20

11. Secondary Outcome: Hospice Consult (Chart Review)
Description: Hospice use for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of hospice use between study arms.
Time Frame: 30 days prior to death
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 26 | 32
Participants | 9 | 16

12. Secondary Outcome: Palliative Care Consult (Chart Review)
Description: Palliative Care consult for each patient will be abstracted by electronic medical record chart review for each patient at 12 months after enrollment. We will evaluate comparisons of palliative care use between study arms.
Time Frame: 6 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
Participants | 37 | 55
Statistical Analysis 1: Comparison: Arm A (Usual Care) vs Arm B (Health Care Coach Support); Test type: Superiority; Odds Ratio (OR) = 4.46, 95% CI 2-sided [1.88 to 10.55]

13. Secondary Outcome: Palliative Care Consult (Chart Review)
Description: as for outcome 12
Time Frame: 12 months after patient enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 64 | 64
Participants | 37 | 55

14. Secondary Outcome: Palliative Care Consult (Chart Review)
Description: Palliative Care consult for each patient will be abstracted by electronic medical record chart review for each patient who has died. We will evaluate comparisons of palliative care use between study arms.
Time Frame: 30 days prior to death
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
Number analyzed (Participants) | 26 | 32
Participants | 17 | 26

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm A (Usual Care) | Arm B (Health Care Coach Support)
All-Cause Mortality (participants affected / at risk) | 26/64 | 32/64
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/64
Other Adverse Events (participants affected / at risk) | 0/64 | 0/64

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/90/NCT03154190/Prot_SAP_000.pdf